CLINICAL TRIAL: NCT06723873
Title: The Immediate Effects of Kinesiology Taping on the Trunk-Scapula-Shoulder Complex in Stroke Patients: A Placebo-Controlled Study
Brief Title: Effects of Kinesiology Taping in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Özge Tahran, Assistant Professor, University of Beykent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108400987-244
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Upper Extremity Dysfunction
Keywords: stroke; trunk control; kinesiology taping
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiology Taping Group (Experimental): Each taping method was carefully designed to address the unique muscle imbalances and functional deficits commonly seen in stroke patients.
  Interventions: Other: Kinesiology Taping
- Placebo-Controlled Sham Group (Sham Comparator): Utilizing three 'I'-shaped strips placed superficially on the skin to ensure no therapeutic effects were achieved.
  Interventions: Other: Placebo Kinesio Taping

INTERVENTIONS:
Other: Kinesiology Taping — The treatment group received Kinesiology Taping around the trunk extensors, lower and middle trapezius, supraspinatus, deltoid muscle group, and serratus anterior muscle.
  Arms: Kinesiology Taping Group
Other: Placebo Kinesio Taping — In the control group, kinesiology tape was applied without tension and in a manner that did not target specific muscle groups or respect the anatomical origin and insertion points.
  Arms: Placebo-Controlled Sham Group

SUMMARY:
The goal of this clinical trial is to learn if kinesiology taping works to treat stroke patients. The main question it aims to answer is:

Is kinesiology taping effective in stroke patients? Researchers compare kinesiology taping to a placebo (visually similar but has no effects) to see if kinesiology taping works immediately to treat stroke patients.

DETAILED DESCRIPTION:
This study aimed to evaluate the immediate effects of kinesiology taping (KT) on trunk control, posture, proprioception, and upper limb function in stroke patients, specifically focusing on the trunk-scapula-shoulder complex. A total of thirty-seven stroke patients participated in this placebo-controlled trial, where they were randomly assigned to either the KT group (n=19) or a placebo-controlled sham KT group (n=18). The KT group received kinesiology taping applied using facilitation and inhibition techniques, while the control group received sham taping without therapeutic tension.

The application of kinesiology taping to the trunk-scapula-shoulder complex in stroke patients resulted in immediate enhancements in trunk control, shoulder posture, and proprioception. However, it did not significantly improve upper limb function in the short term.

ELIGIBILITY:
Inclusion Criteria:

* Experienced a first-ever stroke
* Demonstrated a motor recovery level of Brunnstrom stages 3 or 4 in the affected upper limb
* No history of botulinum toxin-A therapy within the past three months
* Possess sufficient cognitive ability to understand and follow assessment instructions

Exclusion Criteria:

* Individuals with movement or functional limitations due to prior shoulder injuries
* Exhibited allergic reactions or skin sensitivities to taping
* Patients with any existing skin conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
The Trunk Impairment Scale | Change of trunk impairment from baseline at the end of 24 hours of each kinesiology taping intervention.
  The Trunk Impairment Scale (TIS) is a validated assessment tool designed to evaluate trunk function in stroke patients, measuring static sitting balance, dynamic sitting balance, and trunk coordination through a total of 17 items. Each item is scored based on the patient's performance, with the highest score recorded from three repetitions. The TIS provides a total score ranging from 0 to 23 points, where a higher score indicates better trunk function.
Posture Evaluation | Change of posture scores from baseline at the end of 24 hours of each kinesiology taping intervention.
  Posture was assessed using the Posture Screen Mobile (PSM) application, a reliable and valid software tool for posture analysis available on iOS and Android devices. In this study, a physiotherapist utilized an iPad camera to capture sagittal plane photographs of each participant, which were then digitized by marking specific anatomical landmarks. The PSM application calculated anterior and lateral translations, as well as angular displacements, overlaying a grid on the images to assist in accurate landmark placement.
Proprioception Evaluation | Change of proprioception scores from baseline at the end of 24 hours of each kinesiology taping intervention.
  Trunk and shoulder proprioception were evaluated using the inclinometer, with participants positioned at 30° forward flexion of the trunk for testing. They were instructed to hold this position for 5 seconds and then return to a neutral position for another 5 seconds before attempting to reproduce the initial benchmark position, with up to five attempts allowed. Shoulder proprioception was assessed at 75° and 90° flexion.

SECONDARY OUTCOMES:
Motor Assessment Scale | Change of upper-limb function scores from baseline at the end of 24 hours of each kinesiology taping intervention.
  The Motor Assessment Scale (MAS) was employed to evaluate upper-limb function in stroke patients, focusing specifically on three items: item 6 (upper-limb function), item 7 (hand movements), and item 8 (advanced hand activities). Each item is scored on a scale from 0 to 6, with higher scores indicating better functional ability, resulting in a total score range of 0 to 18 for these three items.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Ersöz Hüseyinsinoğlu, Assoc.Prof., Study Director — Marmara University
Locations (1):
- Beykent University, Istanbul, Turkey (Türkiye)